CLINICAL TRIAL: NCT03199924
Title: Intravenous Magnesium Sulfate Combined to Diclofenac Versus Intravenous Lidocaine Combined to Diclofenac Versus Diclofenac Alone in the ED Treatment of Renal Colic. A Randomized Double Blind Study.
Brief Title: Treatment of Renal Colic in the Emergency Departement (ED).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COL-NEPHR
Record Dates: First submitted 2017-05-14; First posted 2017-06-27 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Renal Colic
Keywords: acute pain; Renal colic; Diclofenac; Lidocain; Magnesium sulfate
MeSH Terms: conditions — Renal Colic; Acute Pain | interventions — Diclofenac; Magnesium Sulfate; Lidocaine

STUDY DESIGN:
Intervention Model Description: Double blind study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous Magnesium sulfate combined to Diclofenac (Active Comparator): Intravenous Magnesium sulfate combined to Diclofenac
  Interventions: Drug: Diclofenac; Drug: Magnesium Sulfate
- intravenous lidocaine combined to diclofenac (Active Comparator): intravenous lidocaine combined to diclofenac
  Interventions: Drug: Diclofenac; Drug: Lidocaine
- diclofenac alone (Active Comparator): diclofenac alone
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — Intramuscular injection of 75mg / 3ml of Diclofenac solution
  Other Names: Non Steroidal Anti Inflammatories; Voltaren
Drug: Magnesium Sulfate — intravenous injection of 1 g magnesium solution diluted in 10ml of saline solution administered over 2 minutes
  Other Names: MgSO4; Sulfamag
  Arms: Intravenous Magnesium sulfate combined to Diclofenac
Drug: Lidocaine — intravenous injection of 10ml lidocaine 1% solution administered over 2 minutes
  Other Names: lignocaine; Xylocaine
  Arms: intravenous lidocaine combined to diclofenac

SUMMARY:
to evaluate the analgesic effect of a standard dose of intravenous magnesium added to intramuscular diclofenac compared to intravenous lidocaine combined to intramuscular diclofenac or intramuscular diclofenac alone in patients presenting to the emergency department with renal colic and whether it can reduce opioid consumption.

DETAILED DESCRIPTION:
Magnesium (MgSO4) is a N-Methyl-D-aspartate (NMDA) receptor antagonist and is thought to be involved in the modulation of pain. There has been little direct evidence that MgSO4 relieve neuropathic pain and prevents opioid-induced hyperalgesia in humans.

Intramuscular Diclofenac seems to offer the most effective sustained analgesia for renal colic in the ED and has few side effects.

Lidocain became the agent of choice in visceral and central pain. Intravenous lidocain is effective in the management of neuropathic pain such as diabetic neuropathy, post-surgical pain, post herpetic pain, headaches, and neurological malignancies. At low doses, lidocain is known a relatively safe medication. Lidocain seems an effective treatment who can be administrated in the renal colic.

Objective of study :

The aim of this study is to evaluate the analgesic effect of a standard dose of intravenous magnesium added to intramuscular diclofenac compared to intravenous lidocain combined to intramuscular diclofenac or intramuscular diclofenac alone in patients presenting to the emergency department with renal colic and whether it can reduce opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Age > 18years.
* Confirmed renal colic
* With moderate to severe pain (visual analogic Scale ≥4).

Exclusion Criteria:

* Current regular use of analgesics, anticonvulsants, or antidepressants.
* Analgesia taken within 24 hours .
* Renal disorder with a low glomerular filtration rate (< 60ml/min)
* Neuromuscular disorder.
* Severe cardiac disease.
* Pregnant women
* Contraindication to one of the protocol treatment
* Inability of the patient to cooperate
* Allergy to NSAID or lidocaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Treatment success evaluated at 30 minutes after drug administration. | 30 minutes
  we consider significant pain reduction as a drop in the initial pain score of 50% or more at 30 minutes following analgesia administration.
Pain resolution time evaluated at 5, 10, 30, 60 and 90 minutes after drug administration. | 90 minutes
  elapsed time between the start of the protocol and the decrease of baseline pain score by at least 50%.

SECONDARY OUTCOMES:
The proportion of patients achieving a drop in initial pain score of at least 3 evaluated at 30 minutes | 30 minutes
  The proportion of patients achieving a drop in initial pain score of at least 3
Adverse effect | 90 minutes
  eg nausea, vomiting, vertigo, and lethargy based on self-reports and other clinical manifestations occuring at any moment of the protocol
The need for additional analgesics at 30 minutes after protocol start to relieve the pain | 30 minutes
  The need for rescue analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Nouira semir, professor, Principal Investigator — university of ùmonastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No